CLINICAL TRIAL: NCT06122116
Title: Investigating Orthobiologics After Platelet-Rich Plasma and Photobiomodulation Treatment of Knee Osteoarthritis
Brief Title: Investigating Orthobiologics After PRP and Photobiomodulation for Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Institutional Review Board terminated the protocol on 10 October 2024.
Sponsor: Musculoskeletal Injury Rehabilitation Research for Operational Readiness (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Photomedicine Project 11
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Physical Therapy (PT) Only (Active Comparator): All participants will complete a standard of care PT program addressing individual strength, mobility, and flexibility deficits in both proximal and distal muscle groups. The provider may also use other modalities to address distal issues. If a participant has not been placed on profile at the time of consent, a profile may be written by the study medical provider to ensure limitation of activities, as appropriate.
  Interventions: Other: Physical Therapy
- PT + Platelet-Rich Plasma (PRP) (Active Comparator): PRP Preparation: The PRP will be prepared following standard technique by drawing 60cc blood from the participant through venipuncture and spinning the blood sample in a centrifuge (for approximately 17 minutes), adjusting for leukocyte poor-platelet rich plasma (LP-PRP). This sample will be prepared by the study provider. Any leftover blood will be safely discarded per standard protocols.
  A small portion of the pre-spin whole blood (approximately 1 cc) and post-spin injectant PRP (approximately 1 cc) will be sent to MAMC Department of Pathology and Laboratory Services (DPALS) for complete blood count (CBC) cytology to monitor standardization and reproducibility. This portion will be labeled by participant ID and study. De-identified hardcopy results will be obtained from MAMC DPALS, and CBC results will be reported on Appendix G (CBC Results CRF). Post-procedural instructions will be provided in a participant handout.
  Interventions: Other: Physical Therapy; Biological: Platelet-Rich Plasma Injection
- PT + Photobiomodulation Treatment (PBMT) (Active Comparator): In addition to SOC PT, the PBMT group will receive PBM treatment, as outlined below.
  PBM treatments will occur 3 times each week, for 3 weeks. A member of the study team will measure the treatment area according to a standard protocol and calculate the treatment time (approximately 5-20 minutes). PBMT will be delivered at 6 J/cm2 and 25W and applied in a serpentine pattern to the knee area. Participants will be asked to refrain from using perfumes or plant extracts (e.g., St. John's Wort) in the treatment area(s), as this can increase skin photosensitivity.
  Interventions: Other: Physical Therapy; Device: Photobiomodulation Therapy
- PT + PRP + PBMT (Active Comparator): In addition to SOC PT, the PRP and PBMT group will receive PRP treatment and PBMT treatments.
  Participants in this group will start PBMT treatments on the same day after receiving the study PRP injection. On the day of the PRP injection, the participant will be instructed to rest for 5-10 minutes prior to the PBMT application and team member will ensure the participant is comfortable not in pain. Immediately following the study injection, the team member will take care not to provide the PBMT over the injected area; however, all subsequent PBMT treatments will be delivered to the knee where the PRP was injected.
  Interventions: Other: Physical Therapy; Biological: Platelet-Rich Plasma Injection; Device: Photobiomodulation Therapy

INTERVENTIONS:
Other: Physical Therapy — The PT treatment participants receive in this study will be standard of care; that is, the PT treatment regimen will not be standardized across study participants and/or dictated by study-specific criteria. Participants will be referred to the Physical Therapy Department at the Madigan Army Medical Center (MAMC). Number of PT treatments will be documented on a follow-up Chart Review.
  Other Names: SOC PT
Biological: Platelet-Rich Plasma Injection — PRP injection procedures will follow current clinical recommendation and standard operating procedures. Prior to the injection, the area will be sterilely prepared and anesthetized with either ethyl chloride spray or lidocaine (limited to the cutaneous and subcutaneous layer, so as not to alter the synovial contents). Then, the participant will receive LP-PRP injection in the affected knee area under ultrasound guidance. Qualified study providers will inject 2-5cc LP-PRP using an 18-gauge 1/5-inch needle for both aspiration and subsequent injection. Study providers will select the injection portal they are most comfortable with, in order to achieve an accurate intra-articular injection. The PRP injection procedure is expected to take approximately one hour.
  Other Names: PRP
  Arms: PT + PRP + PBMT; PT + Platelet-Rich Plasma (PRP)
Device: Photobiomodulation Therapy — PBMT is delivered with the LightForce® XPi 25W device through the Smart Hand Piece technology. PBMT will be delivered at 6 J/cm^2 and applied in a circular pattern to the knee area.
  Other Names: PBMT
  Arms: PT + PRP + PBMT; PT + Photobiomodulation Treatment (PBMT)

SUMMARY:
This research assesses the effects that Photobiomodulation Therapy (PBMT) has on Intra-articular administered Plasma-Rich Platelet (PRP) injections for Knee Osteoarthritis (KOA) treatment through evaluations of synovial and serum inflammatory and reparative biomarkers.

A comparison of Physical Therapy (PT) vs PT + PRP vs PT + PBMT vs PT + PRP + PBMT for KOA treatment is made. The relationship between self-reported pain and functionality and treatment mechanisms is analyzed along with an analysis of the intersectionality between participant self-reported pain and functionality and medicine markers across treatment groups. These aims seek to inform current treatment practices in treating KOA and returning Active-Duty Service Members to duty readiness.

DETAILED DESCRIPTION:
Post Traumatic Knee Osteoarthritis (PTOA) is a degenerative joint disease resulting in the loss of cartilage due to wear and tear or by an uncharacteristic force applied to the knee. This disease appears frequently in Active-Duty Service Members and is rising in prominence where over 20,000 Knee Osteoarthritis (KOA) cases were detected over a 10-year period. Current treatments such as physical therapy (PT), braces, oral pain relievers, corticosteroid, and hyaluronic acid injections for KOA only address the quality of life and the symptoms but have not demonstrated a reverse in disease progression. Studies have found that Platelet-Rich Plasma (PRP) has shown to be a promising treatment 6-12 months post procedure and may slow KOA progression.

Photobiomodulation therapy (PBMT) is a non-invasive treatment option shown to reduce pain, increase function, and decrease stiffness with or without therapeutic exercises in KOA patients. In combination, PRP and PBMT may increase the recovery benefits while and potentially reduce KOA progression while seeking therapy. The exact dosage for the optimization of treatment with both PRP and PBMT still needs to be analyzed and understood. Therefore, this study will investigate four treatment arms utilizing PT, PT plus PRP, PT plus PBMT, and PT plus PRP plus PBMT. This discover based and randomized control trial will investigate the effect of PBMT and intra-articular administered PRP treatment on clinical outcomes (e.g., pain scores) and biomolecular signatures (DNA, RNA, or protein levels) in the blood or synovial spaces.The participants' intersectionality between pain, functionality, and precision medicine markers will be analyzed across treatment groups. Follow-up data in the form of questionnaires and activity logs will be collected to monitor study progression.

ELIGIBILITY:
Inclusion Criteria:

* DEERS Eligible
* Between 18-64 (Inclusive)
* Civilian
* Contractor
* Active Duty Service Member
* Knee Osteoarthritis diagnosis

  a) at least 3 of the following:
  1. >50 years old
  2. Morning stiffness < 30 minutes
  3. Crepitus on active movements
  4. Tenderness of the bony margins of the joint
  5. Bony enlargement
  6. No palpable warmth
* Fluent in speaking and reading English
* Ability to commit to study intervention and follow-up
* Willing to avoid prohibited treatments while enrolled in the study (NSAIDs/COX-2 inhibitors and ASAs for 5 days prior to and 2 weeks following study injection or beginning of treatment, and oral steroids, steroid injections, and viscos supplementation)
* Radiographic evidence of knee osteoarthritis as assessed by Kellgren-Lawrence grade 1 or higher

Exclusion Criteria:

* Current participation in other research studies for knee OA
* Previous enrollment for contralateral knee
* Hx of arthroscopic surgery on the study knee within the past year
* Hx of arthroplasty on the study knee
* Received dry needling within the past 4 weeks
* Received prolotherapy (e.g. CSI or PRP injection), within past month
* Recent (within the last 3 months) lower extremity injury (e.g., ankle sprain, meniscus tear or sprain, etc.) that required professional medical attention, and occurred in the ipsilateral extremity of the study knee
* Confounding, coexisting pathology suspected to be the primary source of their pain [e.g., acute meniscal tear (with mechanical symptoms), ligamentous changes (with clinical instability) or hemarthrosis]
* Current or chronic sciatica (lumbosacral radiculopathy) resulting in chronic or intermittent lower extremity pain, numbness, or tingling
* Diagnosis of neuropathy affecting sensation to pain
* Diagnosis of inflammatory arthropathy
* Diagnosis of fibromyalgia or chronic fatigue syndrome
* Hx of adverse reaction to PRP injection (either documented in the medical record or shared by the patient during screening)
* Tattoo in treatment area
* Diagnosis of porphyria (light induced allergy) or photosensitive eczema
* Current use of medications associated with sensitivity to heat or light (e.g., amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
* Current use of pacemaker
* Hx of underlying cardiac disease
* Diagnosis of autoimmune disease
* Albinism
* Current pregnancy or plans to become pregnant during intervention period
* Hx of memory problems, dementia, and/or impaired decision-making ability
* Any other serious medical conditions(s) that might preclude optimal outcome and/or interfere with participation (e.g.), intra-articular sepsis, bacteremia, fracture, joint instability, rheumatoid arthritis, osteoporosis, cancer, coagulopathy, etc.)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Kellgren Lawrence Classification System (KL) | Baseline
  Kellgren Lawrence Classification System (KL) will score the radiographic evidence of the participant's knee osteoarthritis.
  Minimum Score: Grade 0 (none): definite absence of X-ray changes of knee OA
  Maximum Score: Grade 4 (severe): Large osteophyte formation, joint space narrowing, definite bone end deformity
  Higher grades indicate a worse outcome.
Defense and Veterans Pain Rating Scale (DVPRS) | Baseline
  Defense and Veterans Pain Rating Scale (DVPRS) will capture current pain severity.
  Minimum Score: 0 (no pain)
  Maximum Score: 10 (As bad as it could be, nothing else matters)
  A higher score indicates, increasing pain.
Defense and Veterans Pain Rating Scale (DVPRS) | Daily, for 6 weeks
  Defense and Veterans Pain Rating Scale (DVPRS) will capture current pain severity.
  Minimum Score: 0 (no pain)
  Maximum Score: 10 (As bad as it could be, nothing else matters)
  A higher score indicates, increasing pain.
Single Assessment Numeric Evaluation (SANE) | Baseline
  Single Assessment Numeric Evaluation (SANE) will rate the participant's knee osteoarthritis condition as a percentage from normal.
  Minimum Score: 0% (Abnormal)
  Maximum Score: 100% (Fully Normal)
  An increasing percentage means the closer the participant feels their knee is back to normal function.
Single Assessment Numeric Evaluation (SANE) | Daily, for 6 weeks
  Single Assessment Numeric Evaluation (SANE) will rate the participant's knee osteoarthritis condition as a percentage from normal.
  Minimum Score: 0% (Abnormal)
  Maximum Score: 100% (Fully Normal)
  An increasing percentage means the closer the participant feels their knee is back to normal function.
Knee Injury Osteoarthritis Outcome Score (KOOS) | Baseline
  Knee Injury Osteoarthritis Outcome Score (KOOS) will ask the participants questions while thinking about their injured knee symptoms in the past week.
  Minimum Score: None
  Maximum Score: Extreme
  On a per question basis, the participant states how significant their knee symptoms are.
Knee Injury Osteoarthritis Outcome Score (KOOS) | 3-week follow-up
  Knee Injury Osteoarthritis Outcome Score (KOOS) will ask the participants questions while thinking about their injured knee symptoms in the past week.
  Minimum Score: None
  Maximum Score: Extreme
  On a per question basis, the participant states how significant their knee symptoms are.
Knee Injury Osteoarthritis Outcome Score (KOOS) | 6-week follow-up
  Knee Injury Osteoarthritis Outcome Score (KOOS) will ask the participants questions while thinking about their injured knee symptoms in the past week.
  Minimum Score: None
  Maximum Score: Extreme
  On a per question basis, the participant states how significant their knee symptoms are.
The Veterans Rand 12 Item Health Survey (VR-12) | Baseline
  The Veterans Rand 12 Item Health Survey (VR-12) asks participants about their feelings and how well they can do their usual activities.
  Minimum Score 1: Poor Maximum Score 1: Excellent Refers to a participant's general health.
  Minimum Score 2: Yes, limited a lot Maximum Score 2: No, not limited at all Refers to activity, how their health has limited them.
  Minimum Score 3: No, none of the time Maximum Score 3: Yes, all of the time How Physical health has that impacted accomplishments and the kind of work of other activities.
  Minimum Score 4: Not at all Maximum Score 4: Extremely Refers to how pain interferes with normal work.
  Minimum Score 5: All of the time Maximum Score 5: None of the time Refers to feeling calm, having energy, and whether they feel downhearted.
  Minimum Score 6: Much worse Maximum Score 6: Much better A comparison of physical health compared to a year ago and a comparison of emotional health compared to a year ago.
The Veterans Rand 12 Item Health Survey (VR-12) | 3-week follow-up
  The Veterans Rand 12 Item Health Survey (VR-12) will ask participants about how they feel and how well they are able to do their usual activities.
  Minimum Score 1: Poor Maximum Score 1: Excellent Refers to a participant's general health.
  Minimum Score 2: Yes, limited a lot Maximum Score 2: No, not limited at all Refers to activity, how their health has limited them.
  Minimum Score 3: No, none of the time Maximum Score 3: Yes, all of the time How Physical health has that impacted accomplishments and the kind of work of other activities.
  Minimum Score 4: Not at all Maximum Score 4: Extremely Refers to how pain interferes with normal work.
  Minimum Score 5: All of the time Maximum Score 5: None of the time Refers to feeling calm, having energy, and whether they feel downhearted.
  Minimum Score 6: Much worse Maximum Score 6: Much better A comparison of physical health compared to a year ago and a comparison of emotional health compared to a year ago.
The Veterans Rand 12 Item Health Survey (VR-12) | 6-week follow-up
  The Veterans Rand 12 Item Health Survey (VR-12) will ask participants about how they feel and how well they are able to do their usual activities.
  Minimum Score 1: Poor Maximum Score 1: Excellent Refers to a participant's general health.
  Minimum Score 2: Yes, limited a lot Maximum Score 2: No, not limited at all Refers to activity, how their health has limited them.
  Minimum Score 3: No, none of the time Maximum Score 3: Yes, all of the time How Physical health has that impacted accomplishments and the kind of work of other activities.
  Minimum Score 4: Not at all Maximum Score 4: Extremely Refers to how pain interferes with normal work.
  Minimum Score 5: All of the time Maximum Score 5: None of the time Refers to feeling calm, having energy, and whether they feel downhearted.
  Minimum Score 6: Much worse Maximum Score 6: Much better A comparison of physical health compared to a year ago and a comparison of emotional health compared to a year ago.
Biorepository Blood Draw for Biomarkers of Interest ADAMTS-4 &5 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: ADAMTS-4 &5.
Biorepository Blood Draw for Biomarkers of Interest MMP 7 & 9 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: MMP 7 & 9.
Biorepository Blood Draw for Biomarkers of Interest TGF-B | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: TGF-B.
Biorepository Blood Draw for Biomarkers of Interest Aggrecan | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: Aggrecan.
Biorepository Blood Draw for Biomarkers of Interest HYAL2 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HYAL2.
Biorepository Blood Draw for Biomarkers of Interest CRP | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CRP.
Biorepository Blood Draw for Biomarkers of Interest HA | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HA.
Biorepository Blood Draw for Biomarkers of Interest CD14 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD14.
Biorepository Blood Draw for Biomarkers of Interest CD16 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD16.
Biorepository Blood Draw for Biomarkers of Interest CD64 | Baseline
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD64.
Knee Joint Aspiration for Biomarkers of Interest CD64 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD64.
Knee Joint Aspiration for Biomarkers of Interest CD16 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD16.
Knee Joint Aspiration for Biomarkers of Interest CD14 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD14.
Knee Joint Aspiration for Biomarkers of Interest HA | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HA.
Knee Joint Aspiration for Biomarkers of Interest CRP | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CRP.
Knee Joint Aspiration for Biomarkers of Interest HYAL2 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HYAL2.
Knee Joint Aspiration for Biomarkers of Interest Aggrecan | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: Aggrecan.
Knee Joint Aspiration for Biomarkers of Interest TGF-B | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: Aggrecan.
Knee Joint Aspiration for Biomarkers of Interest MMP 7 & 9 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: MMP 7& 9.
Knee Joint Aspiration for Biomarkers of Interest ADAMTS-4 & 5 | Baseline
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: ADAMTS-4 & 5.
Biorepository Blood Draw for Biomarkers of Interest CD64. | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD64.
Biorepository Blood Draw for Biomarkers of Interest CD16 | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD16.
Biorepository Blood Draw for Biomarkers of Interest CD14 | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD14.
Biorepository Blood Draw for Biomarkers of Interest HA | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HA.
Biorepository Blood Draw for Biomarkers of Interest CRP | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CRP.
Biorepository Blood Draw for Biomarkers of Interest HYAL2 | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HYAL2.
Biorepository Blood Draw for Biomarkers of Interest Aggrecan | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: Aggrecan.
Biorepository Blood Draw for Biomarkers of Interest TGF-B | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: TGF-B.
Biorepository Blood Draw for Biomarkers of Interest MMP 7 & 9 | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: MMP 7 & 9.
Biorepository Blood Draw for Biomarkers of Interest ADAMTS-4 & 5 | 6-week follow-up
  4 ml of blood collected in K2/EDTA tube, 4 ml of blood collected in heparin tube, 3 ml of blood collected in DNA/RNA tube. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: ADAMTS-4 & 5.
Knee Joint Aspiration for Biomarkers of Interest ADAMTS-4 & 5 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: ADAMTS-4 & 5.
Knee Joint Aspiration for Biomarkers of Interest MMP 7 & 9 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: MMP 7 & 9.
Knee Joint Aspiration for Biomarkers of Interest TGF-B | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: TGF-B.
Knee Joint Aspiration for Biomarkers of Interest Aggrecan | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: Aggrecan.
Knee Joint Aspiration for Biomarkers of Interest HYAL2 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HYAL2.
Knee Joint Aspiration for Biomarkers of Interest CRP | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CRP.
Knee Joint Aspiration for Biomarkers of Interest HA | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: HA.
Knee Joint Aspiration for Biomarkers of Interest CD14 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD14.
Knee Joint Aspiration for Biomarkers of Interest CD16 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD16.
Knee Joint Aspiration for Biomarkers of Interest CD64 | 6-week follow-up
  Synovial fluid from the knee will be extracted and stored in the biorepository. Once sufficient sampling has been met, batch analyses will be completed for biomarker capture including: CD64.
Complete Blood Count (CBC) Analysis WBC | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of WBC.
Complete Blood Count (CBC) Analysis RBC | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of RBC.
Complete Blood Count (CBC) Analysis HGB | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of HGB.
Complete Blood Count (CBC) Analysis HCT | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of HCT.
Complete Blood Count (CBC) Analysis PLT | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of PLT.
Complete Blood Count (CBC) Analysis LYM% | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of LYM%.
Complete Blood Count (CBC) Analysis LYM# | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of LYM#.
Complete Blood Count (CBC) Analysis MON% | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of MON%.
Complete Blood Count (CBC) Analysis GRA% | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of GRA%.
Complete Blood Count (CBC) Analysis Neutrophil% | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of Neutrophil%.
Complete Blood Count (CBC) Analysis Eosinophil%, | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of Eosinophil%.
Complete Blood Count (CBC) Analysis Basophil% | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of Basophil%.
Complete Blood Count (CBC) Analysis MON# | Baseline
  Whole blood and PRP spin analysis will be completed to analyze total blood content of MON#.

CONTACTS AND LOCATIONS:
Overall Officials: Scott P Grogan, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnoczky SP, Sheibani-Rad S. The basic science of platelet-rich plasma (PRP): what clinicians need to know. Sports Med Arthrosc Rev. 2013 Dec;21(4):180-5. doi: 10.1097/JSA.0b013e3182999712. PMID 24212364
- [Background] Assis L, Milares LP, Almeida T, Tim C, Magri A, Fernandes KR, Medalha C, Renno AC. Aerobic exercise training and low-level laser therapy modulate inflammatory response and degenerative process in an experimental model of knee osteoarthritis in rats. Osteoarthritis Cartilage. 2016 Jan;24(1):169-77. doi: 10.1016/j.joca.2015.07.020. Epub 2015 Aug 5. PMID 26254236
- [Background] Blank ML, Cress EA, Snyder F. Separation and quantitation of phospholipid subclasses as their diradylglycerobenzoate derivatives by normal-phase high-performance liquid chromatography. J Chromatogr. 1987 Apr 17;392:421-5. doi: 10.1016/s0021-9673(01)94286-4. No abstract available. PMID 3597586
- [Background] Cook CS, Smith PA. Clinical Update: Why PRP Should Be Your First Choice for Injection Therapy in Treating Osteoarthritis of the Knee. Curr Rev Musculoskelet Med. 2018 Dec;11(4):583-592. doi: 10.1007/s12178-018-9524-x. PMID 30350299
- [Background] Dhillon MS, Patel S, John R. PRP in OA knee - update, current confusions and future options. SICOT J. 2017;3:27. doi: 10.1051/sicotj/2017004. Epub 2017 Mar 22. PMID 28322719
- [Background] Dompe C, Moncrieff L, Matys J, Grzech-Lesniak K, Kocherova I, Bryja A, Bruska M, Dominiak M, Mozdziak P, Skiba THI, Shibli JA, Angelova Volponi A, Kempisty B, Dyszkiewicz-Konwinska M. Photobiomodulation-Underlying Mechanism and Clinical Applications. J Clin Med. 2020 Jun 3;9(6):1724. doi: 10.3390/jcm9061724. PMID 32503238
- [Background] Filardo G, Previtali D, Napoli F, Candrian C, Zaffagnini S, Grassi A. PRP Injections for the Treatment of Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Trials. Cartilage. 2021 Dec;13(1_suppl):364S-375S. doi: 10.1177/1947603520931170. Epub 2020 Jun 19. PMID 32551947
- [Background] Goncalves AB, Bovo JL, Gomes BS, Pigoso AA, Felonato M, Esquisatto MAM, Filho GJL, do Bomfim FRC. Photobiomodulation (lambda=808nm) and Platelet-Rich Plasma (PRP) for the Treatment of Acute Rheumatoid Arthritis in Wistar Rats. J Lasers Med Sci. 2021 Oct 18;12:e60. doi: 10.34172/jlms.2021.60. eCollection 2021. PMID 35155145
- [Background] Hamblin M, Demidova-Rice TN. Cellular chromophores and signaling in low level light therapy. In Biomedical Optics 2007
- [Background] Hsu H, Siwiec RM. Knee Osteoarthritis. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507884/ PMID 29939661
- [Background] Huang G, Hua S, Yang T, Ma J, Yu W, Chen X. Platelet-rich plasma shows beneficial effects for patients with knee osteoarthritis by suppressing inflammatory factors. Exp Ther Med. 2018 Mar;15(3):3096-3102. doi: 10.3892/etm.2018.5794. Epub 2018 Jan 24. PMID 29599843
- [Background] Ip D. Does addition of low-level laser therapy (LLLT) in conservative care of knee arthritis successfully postpone the need for joint replacement? Lasers Med Sci. 2015 Dec;30(9):2335-9. doi: 10.1007/s10103-015-1814-6. Epub 2015 Sep 29. PMID 26420240
- [Background] Migliorini F, Driessen A, Quack V, Sippel N, Cooper B, Mansy YE, Tingart M, Eschweiler J. Comparison between intra-articular infiltrations of placebo, steroids, hyaluronic and PRP for knee osteoarthritis: a Bayesian network meta-analysis. Arch Orthop Trauma Surg. 2021 Sep;141(9):1473-1490. doi: 10.1007/s00402-020-03551-y. Epub 2020 Jul 28. PMID 32725315
- [Background] Molloy JM, Pendergrass TL, Lee IE, Chervak MC, Hauret KG, Rhon DI. Musculoskeletal Injuries and United States Army Readiness Part I: Overview of Injuries and their Strategic Impact. Mil Med. 2020 Sep 18;185(9-10):e1461-e1471. doi: 10.1093/milmed/usaa027. PMID 32175566
- [Background] Ng NT, Heesch KC, Brown WJ. Strategies for managing osteoarthritis. Int J Behav Med. 2012 Sep;19(3):298-307. doi: 10.1007/s12529-011-9168-3. PMID 21614451
- [Background] O'Connell B, Wragg NM, Wilson SL. The use of PRP injections in the management of knee osteoarthritis. Cell Tissue Res. 2019 May;376(2):143-152. doi: 10.1007/s00441-019-02996-x. Epub 2019 Feb 13. PMID 30758709
- [Background] Paolillo FR, Paolillo AR, Joao JP, Frasca D, Duchene M, Joao HA, Bagnato VS. Ultrasound plus low-level laser therapy for knee osteoarthritis rehabilitation: a randomized, placebo-controlled trial. Rheumatol Int. 2018 May;38(5):785-793. doi: 10.1007/s00296-018-4000-x. Epub 2018 Feb 26. PMID 29480363
- [Background] Peplow PV, Chung TY, Ryan B, Baxter GD. Laser photobiomodulation of gene expression and release of growth factors and cytokines from cells in culture: a review of human and animal studies. Photomed Laser Surg. 2011 May;29(5):285-304. doi: 10.1089/pho.2010.2846. Epub 2011 Feb 10. PMID 21309703
- [Background] Rayegani SM, Raeissadat SA, Heidari S, Moradi-Joo M. Safety and Effectiveness of Low-Level Laser Therapy in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. J Lasers Med Sci. 2017 Summer;8(Suppl 1):S12-S19. doi: 10.15171/jlms.2017.s3. Epub 2017 Aug 29. PMID 29071029
- [Background] Showery JE, Kusnezov NA, Dunn JC, Bader JO, Belmont PJ Jr, Waterman BR. The Rising Incidence of Degenerative and Posttraumatic Osteoarthritis of the Knee in the United States Military. J Arthroplasty. 2016 Oct;31(10):2108-14. doi: 10.1016/j.arth.2016.03.026. Epub 2016 Mar 21. PMID 27181491
- [Background] Stausholm MB, Naterstad IF, Joensen J, Lopes-Martins RAB, Saebo H, Lund H, Fersum KV, Bjordal JM. Efficacy of low-level laser therapy on pain and disability in knee osteoarthritis: systematic review and meta-analysis of randomised placebo-controlled trials. BMJ Open. 2019 Oct 28;9(10):e031142. doi: 10.1136/bmjopen-2019-031142. PMID 31662383
- [Background] Tomazoni SS, Leal-Junior EC, Frigo L, Pallotta RC, Teixeira S, de Almeida P, Bjordal JM, Lopes-Martins RA. Isolated and combined effects of photobiomodulation therapy, topical nonsteroidal anti-inflammatory drugs, and physical activity in the treatment of osteoarthritis induced by papain. J Biomed Opt. 2016 Oct 1;21(10):108001. doi: 10.1117/1.JBO.21.10.108001. PMID 27752702
- [Background] Tomazoni SS, Leal-Junior EC, Pallotta RC, Teixeira S, de Almeida P, Lopes-Martins RA. Effects of photobiomodulation therapy, pharmacological therapy, and physical exercise as single and/or combined treatment on the inflammatory response induced by experimental osteoarthritis. Lasers Med Sci. 2017 Jan;32(1):101-108. doi: 10.1007/s10103-016-2091-8. Epub 2016 Oct 10. PMID 27726040
- [Background] Vassao PG, Parisi J, Penha TFC, Balao AB, Renno ACM, Avila MA. Association of photobiomodulation therapy (PBMT) and exercises programs in pain and functional capacity of patients with knee osteoarthritis (KOA): a systematic review of randomized trials. Lasers Med Sci. 2021 Sep;36(7):1341-1353. doi: 10.1007/s10103-020-03223-8. Epub 2021 Jan 3. PMID 33392780
- [Background] Xiang A, Deng H, Cheng K, Liu H, Lin L, Qu X, Liu S, Shen X. Laser photobiomodulation for cartilage defect in animal models of knee osteoarthritis: a systematic review and meta-analysis. Lasers Med Sci. 2020 Jun;35(4):789-796. doi: 10.1007/s10103-019-02937-8. Epub 2019 Dec 17. PMID 31845042
- [Background] Assis, L, Tim, C, Martignago, C, Rodrigues Gonçalves, S, Muniz Renno, AC. Effectiveness of photobiomodulation therapy and aerobic exercise training on articular cartilage in an experimental model of osteoarthritis in rats. Proceedings of SPIE, Light-Based Diagnosis and Treatment of Infectious Diseases. 2018;10479. https://doi.org/10.1117.12.2291227

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT06122116/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT06122116/ICF_001.pdf